CLINICAL TRIAL: NCT01705041
Title: Preliminary Field Evaluation of a Point-of-Care Transaminase Test
Brief Title: Preliminary Evaluation of a Point-Of-Care Liver Function Test
Acronym: DFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DFA LFT Study
Record Dates: First submitted 2012-08-21; First posted 2012-10-12 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: HIV; Tuberculosis; Drug-Induced Liver Injury
MeSH Terms: conditions — Tuberculosis; Chemical and Drug Induced Liver Injury | interventions — Liver Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostics for All liver function test (LFT) (Experimental): HIV clinic patients meeting targeted enrollment criteria will give fingerstick blood for use on investigational LFT in comparison to routine transaminase test performed at the clinic lab (gold standard)
  Interventions: Device: Diagnostics for All liver function test (LFT)

INTERVENTIONS:
Device: Diagnostics for All liver function test (LFT) — HIV clinic patients meeting targeted enrollment criteria will give fingerstick blood for use on investigational LFT in comparison to routine transaminase test performed at the clinic lab (gold standard)
  Other Names: Diagnostics for All (DFA) liver function test (LFT); ALT; transaminase

SUMMARY:
The proposed preliminary field evaluation will compare a point-of-care (POC) transaminase test with the standard of care test used in an HIV clinic at the Hospital for Tropical Diseases in Ho Chi Minh City, Vietnam.

DETAILED DESCRIPTION:
The DFA transaminase test provides rapid categorical measurement of ALT in a whole blood specimen taken via finger-stick. The test is based on the platform technology of "paper microfluidics" (also known as "patterned paper"), in which hydrophobic barriers are patterned into a sheet of paper in order to create microfluidic, hydrophilic paths within the paper, through which flow can be directed towards specific detection zones. The test is designed for visual color-coded readout in three ALT ranges ("bins") that correspond to the ranges of AST and ALT (<3x the upper limit of normal (ULN), 3-5x ULN, and >5x ULN) currently used for clinical management decisions per US TB and HIV treatment guidelines. The bin cutoffs are common to treatment guidelines used around the globe, including those used by the Vietnam Ministry of Health.

The colorimetric readout is designed to be read by eye using a visual "read guide" allowing the reader to make a semi-quantitative estimate or assign a categorical value into one of three bins. Alternatively, if the device is scanned (e.g. desk-top scanner) or photographed (e.g. cell phone or standard digital camera, see (9)) and read with image-analysis software, it should be possible to generate a quantitative result. Additionally, multiple control zones notify the user of insufficient sample volume, hemolysis, or damaged reagents.

The overall goal of this study is to conduct a preliminary field evaluation of an investigational transaminase test in a population at risk for DILI. The primary objectives are:

1. Determine device accuracy by measuring the percent agreement of the categorical visual readout DFA transaminase test and the standard of care tests used in the HTD HIV clinic.
2. Determine inter-operator variability.
3. Determine device failure rate as defined by invalid test results.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) patients receiving HIV treatment through the HTD clinic
* Must be receiving routine scheduled ALT monitoring on day of enrollment
* Willing to undergo finger-stick in addition to routine care
* Must be able to provide informed consent.

Exclusion Criteria:

* HIV-negative, or HIV-positive but not on treatment
* Not receiving transaminase monitoring for routine care
* Unable or unwilling to provide informed consent
* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
percent agreement with gold standard test | at time of draw
  Determine device accuracy by measuring the percent agreement of the categorical visual readout DFA transaminase test and the standard of care tests used in the HTD HIV clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Nira Pollock, MD,PhD, Principal Investigator — Harvard University
Locations (1):
- Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam